CLINICAL TRIAL: NCT07271342
Title: Observational Registry of Effectiveness and Safety of Tenecteplase in Real World Settings in China-ORIENTAL
Brief Title: Observational RegIstry of Effectiveness and Safety of teNecTeplase in reAl worLd Settings in China
Acronym: ORIENTAL
Status: Recruiting | Type: Observational
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Yongjun Wang, professor, Beijing Tiantan Hospital
Other Study IDs: CSA2025KY002
Record Dates: First submitted 2025-11-28; First posted 2025-12-09 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Stroke
Keywords: ischemic stroke; tenecteplase; registry
MeSH Terms: conditions — Stroke; Ischemic Stroke | interventions — Tenecteplase

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Tenecteplase-Treated AIS Cohort
  Interventions: Drug: tenecteplase

INTERVENTIONS:
Drug: tenecteplase — Intravenous administration of tenecteplase at a single weight-based dose of 0.25 mg/kg (maximum 25 mg), delivered as an intravenous bolus over 5-10 seconds as part of routine clinical care for acute ischemic stroke. Tenecteplase is used as the sole thrombolytic agent in this observational cohort and is not compared against alteplase or any other active control.

SUMMARY:
The ORIENTAL study is a prospective, multicenter, continuously enrolled real-world cohort designed to evaluate the effectiveness and safety of intravenous tenecteplase for acute ischemic stroke (AIS) in routine clinical practice across China. Approximately 10,000 patients from about 200 hospitals will be included. Eligible adults with imaging-confirmed AIS who receive tenecteplase as part of standard care will be consecutively enrolled and followed through 90 days. The study will describe patient characteristics, treatment processes, functional outcomes, and safety events, and will also explore inter-hospital variability and subgroup differences to support quality improvement and guide nationwide implementation of tenecteplase therapy.

DETAILED DESCRIPTION:
This real-world observational registry aims to generate comprehensive and high-quality evidence on the use of intravenous tenecteplase for acute ischemic stroke (AIS) in China following the national approval of the drug. Unlike randomized controlled trials with strict eligibility criteria, this study captures a broad clinical spectrum of patients and care settings, reflecting the actual patterns, challenges, and variations in stroke management across the country.

The registry is designed to provide insights into how tenecteplase performs in routine practice, including patients with multiple comorbidities, diverse stroke etiologies, and differing hospital capabilities. Consecutive enrollment and continuous data capture ensure representativeness and minimize selection bias.

Beyond describing effectiveness and safety, the study evaluates the real-world processes surrounding thrombolysis, including workflow metrics such as door-to-needle time and access to reperfusion resources. Analyses across different regions, hospital levels, and clinical subgroups will help identify practice gaps and opportunities for nationwide quality improvement. Comparisons with previous phase III trial populations, including the ORIGINAL study, will allow assessment of potential channeling bias and help interpret differences between clinical trial efficacy and real-world effectiveness.

The results of this registry will support clinical decision-making, inform guideline updates, and contribute to establishing standardized stroke care pathways for tenecteplase in China. The large sample size and national coverage are intended to ensure sufficient precision for outcome estimation and enable robust exploratory analyses that can guide future research and policy development.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 18 years or older;
2. Diagnosed with acute ischemic stroke confirmed by imaging (CT or MRI);
3. Treated with intravenous tenecteplase at the participating institution;
4. Provided written informed consent, signed by the patient or their legally authorized representative;
5. Capable of completing follow-up assessments.

Exclusion Criteria:

1. Received reperfusion therapy prior to the hospital admission (e.g., intravenous thrombolysis prior to admission);
2. Participating in any clinical trials where the intervention may affect the outcomes of this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults diagnosed with acute ischemic stroke who receive intravenous tenecteplase as part of routine clinical care at participating hospitals across China. The study population reflects a broad real-world stroke population, including patients with diverse comorbidities, stroke severities, and treatment pathways. Consecutive enrollment from approximately 200 centers ensures representative coverage of different geographic regions and hospital levels.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2025-11-30 (Actual); Primary Completion 2029-03-31 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Favorable functional outcome at 90 days (modified Rankin Scale [mRS] score ≤1) | 90 days

SECONDARY OUTCOMES:
Functional independence at 90 days (mRS score of 0-2) | 90 days
Ordinal mRS score at 90 days | 90 days
Change in NIHSS score at 24 hours compared to baseline (short-term outcome) | 24 hours
Change in NIHSS score at day 7 or discharge compared to baseline (short-term outcome) | 7 days
Symptomatic intracranial hemorrhage (sICH) within 36 hours after intravenous thrombolysis | 36 hours
All-cause mortality and time to death within 90 days | 90 days
Stroke recurrence and time to recurrence within 90 days | 90 days
Serious adverse events during hospitalization | 7days

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tiantan Hospital, Capital Medical University, Beijing, China